CLINICAL TRIAL: NCT02087852
Title: Kidney Cancer DNA Registry
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-218
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Renal Cancer
Keywords: Questionnaire; DNA; saliva; kidney cancer; 13-218; high risk
MeSH Terms: conditions — Kidney Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva specimen
  blood
  tissue (when available)

GROUPS / COHORTS (4):
- kidney cancer patients receiving care at MSKCC: Participation will consist of completing the Kidney Cancer Questionnaire Family History Questionnaire and complete the Epidemiologic Questionnaire (when applicable,), and providing a blood sample and saliva sample for germline DNA. In cases where tissue samples from surgically derived tumor specimens are obtained these will used to determine genetic alterations related to cancer predisposition or pathogenicity.
  Interventions: Other: salvia for germline DNA; Behavioral: the Kidney Cancer Questionnaire; Behavioral: Family History Questionnaire (when applicable); Other: Blood draw; Behavioral: Epidemiologic Questionnaire
- relatives of patients with kidney cancer: Participation will consist of completing the Kidney Cancer Questionnaire Family History Questionnaire (when applicable,), and providing a saliva sample for germline DNA. In cases where tissue samples from surgically derived tumor specimens are obtained these will used to determine genetic alterations related to cancer predisposition or pathogenicity.
  Interventions: Other: salvia for germline DNA; Behavioral: the Kidney Cancer Questionnaire; Behavioral: Family History Questionnaire (when applicable)
- healthy controls who are unrelated & do not have hx of cancer: Participation will consist of completing the Kidney Cancer Questionnaire Family History Questionnaire (when applicable,), and providing a saliva sample for germline DNA. In cases where tissue samples from surgically derived tumor specimens are obtained these will used to determine genetic alterations related to cancer predisposition or pathogenicity.
  Interventions: Other: salvia for germline DNA; Behavioral: the Kidney Cancer Questionnaire; Behavioral: Family History Questionnaire (when applicable)
- high risk: Participation will consist of completing the Epidemiologic Questionnaire, Family History Questionnaire (if + FH), provide saliva and blood sample , referral for screening evaluation
  Interventions: Other: salvia for germline DNA; Behavioral: Family History Questionnaire (when applicable); Other: Blood draw; Behavioral: Epidemiologic Questionnaire

INTERVENTIONS:
Other: salvia for germline DNA
Behavioral: the Kidney Cancer Questionnaire — Patients will complete the appropriate surveys on either paper or on the computer/iPad in the office using REDCap software. If patients are unable to complete their questionnaires at the time of their in-office visit, a link to the questionnaires in REDCap will be emailed to them. The survey data that is collected in REDCap will be stored in REDCap. Clinic staff may also call patients to remind patients to complete questionnaires.
  Groups: healthy controls who are unrelated & do not have hx of cancer; kidney cancer patients receiving care at MSKCC; relatives of patients with kidney cancer
Behavioral: Family History Questionnaire (when applicable) — Patients will complete the appropriate surveys on either paper or on the computer/iPad in the office using REDCap software. If patients are unable to complete their questionnaires at the time of their in-office visit, a link to the questionnaires in REDCap will be emailed to them. The survey data that is collected in REDCap will be stored in REDCap. Clinic staff may also call patients to remind patients to complete questionnaires.
Other: Blood draw
  Groups: high risk; kidney cancer patients receiving care at MSKCC
Behavioral: Epidemiologic Questionnaire — Patients will complete the appropriate surveys on either paper or on the computer/iPad in the office using REDCap software. If patients are unable to complete their questionnaires at the time of their in-office visit, a link to the questionnaires in REDCap will be emailed to them. The survey data that is collected in REDCap will be stored in REDCap. Clinic staff may also call patients to remind patients to complete questionnaires.
  Groups: high risk; kidney cancer patients receiving care at MSKCC

SUMMARY:
This registry will help us develop better methods of:

* Preventing these cancers
* Diagnosing these cancers
* Treating these cancers

ELIGIBILITY:
Inclusion Criteria:

Kidney Cancer Case Cohort:

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must have a diagnosis or suspicion of kidney cancer

Family Member Cohort:

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must be a blood relative of the proband. Family members of probands including mother, father, sisters, brothers, half-sisters, half-brothers, daughters, sons, grandmothers, grandfathers, as well as aunts and uncles are eligible. These individuals need not have kidney cancer, as they will be used for segregation analysis of suspected variants found in the proband; requesting DNA from relatives is required.

Control Cohort:

* Must be ≥ 18 years of age AND
* Must be an English-speaker AND
* Must not have a personal history of cancer, with the exception of nonmelanoma skin cancer, AND
* Must not be a blood relative of any cases or controls enrolled in this study

Exclusion Criteria:

* Patients who, in the opinion of the primary MSKCC clinician or the investigator, have a condition that precludes their ability to provide an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urologists, clinical geneticists, and medical oncologists at MSKCC, along with study personnel will identify patients, family members, and unaffected controls that may be eligible for the registry. Patients and families may also be directly referred to the MSKCC study team by any MSKCC physician, external physician, or by the family itself.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2014-03; Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
establish a kidney cancer registry | 5 years
  with detailed epidemiologic data and germline DNA available for next generation sequencing from consenting patients, selected family members, and healthy unrelated controls.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jonathan, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Consent and Follow-up), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and Follow up), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow up ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-up), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow up), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/